CLINICAL TRIAL: NCT03689036
Title: Transmission Dynamics of Residual and Re-emerging Malaria in the Amazon: Defining a Roadmap to Malaria Elimination_Part A: Acre, Brazil
Brief Title: Transmission Dynamics of Residual and Re-emerging Malaria in the Amazon: Defining a Roadmap to Malaria Elimination
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Simone Ladeia, Investigator, Oswaldo Cruz Foundation
Other Study IDs: DMID 17-0037-A
Record Dates: First submitted 2018-09-25; First posted 2018-09-28 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Malaria
Keywords: malaria; transmission; Asymptomatic infeccion; malaria elimination; residual malaria; Amazon
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasmodium vivax and Plasmodium falciparum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A population baseline longitudinal study in a major residual malaria hotspot in Brazil to: 1. identify risk factors for residual malaria infection and disease at individual and household level, 2. identify and quantify population changes in P. vivax and P. falciparum to detect reintroductions and to estimate parasite population complexity at baseline and after interventions and 3. describe changing dynamics of malaria incidence and parasitemia prevalence over time, and to assess potential effects of combinations of interventions on malaria control and elimination using mathematical models.

The study will be developed in Mâncio Lima, a residual malaria hotspot in northwestern Brazil. The population of study is approximately 2,000 subjects aged 3 months and up, who correspond to all the residents of 20% of the households of the urban area of Mâncio Lima.

Will be made Active (ACD) and Passive Case Detection (PCD) every 6 months, over 5 years. (symptom based surveying; microscopy-based diagnosis).

Each visit will include interview, physical examination and collection of 100 μL of blood (finger prick) to malaria diagnosis by smear, RDT and qPCR. If the subject will be positive by smear or RDT (rapid diagnostic test for malaria), despite of presence of symptoms, ≥ 20 mL of venous blood will be draw of them to immunology and parasite genetics study and the immediate treatment per MOH(Ministry of Health) guidelines will be performed.

Subjects with smear or RDT negative, will be followed for symptoms over the next 6 months. If it is subsequently found to be smear/RDT-positive by PCD, the treatment will be performed.

Clinical and epidemiological characteristics of malaria, genetic characteristics of the population of Plasmodium and changing dynamics of malaria transmission will be analyzed.

DETAILED DESCRIPTION:
Cross-sectional surveys will be carried out in order to identify risk factors for residual malaria infection and disease at both the individual and household level, to supply parasite samples for detailed population-level molecular analyses and to supply epidemiological data for parameterization of new mathematical models of malaria transmission.

SPECIFIC AIMS:

* Aim 1: Longitudinally determine malaria dynamics in a major residual malaria hotspot in Brazil.
* Aim 2: Identify and quantify population changes in P. vivax and P. falciparum to detect reintroductions, and to estimate parasite population complexity at baseline and potentially after interventions.
* Aim 3: Develop and apply mathematical models to describe changing dynamics of malaria incidence and parasitemia prevalence over time, and to assess potential effects of combinations of interventions on malaria control and elimination.

  * The study will be developed in the urban area of Mâncio Lima, northwestern of Brazil.

A census performed by our field team between Nov 2015 and Apr 2016 identified ~ 10,000 inhabitants in the urban area of Mâncio Lima. At the site preparation phase, a random sample of 20% of the households enumerated during our census will be visited by our field teams and all dwellers aged 3 months or up (or their parents/guardians) will be invited to participate in the cohort study.

We expect to enroll ~ 2,000 subjects who will participate in 10 cross-sectional surveys (every six months) over five years (total of 20,000 observations), and contribute 120,000 person-months of follow-up. Because of the open-cohort design of this study, subjects who are lost for follow-up are replaced with newcomers, without affecting significantly the number of person-months of follow-up.

At each visit, the subjects will be interviewed and 100ul of blood will be collected to Active (ACD) and Passive Case Detection (PCD) (symptom based surveying; microscopy-based diagnosis). Each visit will include an interview, physical examination and collection of 100 μL of blood (finger prick) to malaria diagnosis by smear, RDT and qPCR.

When the subjects are positive by smear or RDT (rapid diagnostic test for malaria), despite of presence of symptoms, ≥ 20 mL of venous blood will be draw of them to immunology and parasite genetics study and the immediate treatment per Ministry of Health of Brazil guidelines will be performed.

ELIGIBILITY:
INCLUSION CRITERIA:

* Any subject aged 3 or more months old living in the study sites and providing written informed consent, or with parental written informed consent and assent when age-appropriate;
* Plans to remain in the study site for the next five years.

Adults and children will both contribute to the data and study goals. Adults and children will both contribute to the data and study goals. Children less than three months of age will be excluded from the study because the heel or finger prick procedures to draw blood may be perceived by the parents as inappropriate for this age group. Children aged three months or more are eligible as long as they are members of the randomly chosen households and their parents/guardians provide informed consent. Inclusion of children is essential for the study goals, since different age groups may differ in acquired immunity and therefore in the risk of having symptoms when carrying malaria parasites

EXCLUSION CRITERIA:

* any chronic or acute condition that, in the opinion of the field clinician or nurse, may affect the results of the study or the ability of providing informed consent.
* Less then 3 months old
* Do not have permanent residence in the study area

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A census performed by our field team between Nov 2015 and Apr 2016 identified ~ 10,000 inhabitants in the urban area of Mâncio Lima. At the site preparation phase, a random sample of 20% of the households enumerated during our census will be visited by our field teams and all dwellers aged 3 months or up (or their parents/guardians) will be invited to participate in the cohort study. We expect to enroll ~ 2,000 subjects who will participate in 10 cross-sectional surveys over five years (total of 20,000 observations), and contribute 120,000 person-months of follow-up. Because of the open-cohort design of this study, subjects who are lost for follow-up are replaced with newcomers, without affecting significantly the number of person-months of follow-up.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-04-02 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Risk factors for residual malaria infection and disease | 2023
  Determining sociodemographic variables that are significantly associated with malaria infection (regardless of symptoms) and clinical illness by multilevel multiple regression analysis

SECONDARY OUTCOMES:
Genetic characterization of locally circulating malaria parasites over space and time | 2023
  Determination of multilocus genotypes (using microsatellite markers) and complete genomes of Plasmodium vivax and Plasmodium falciparum isolates obtained from georeferenced households over the study period (5 years).
Estimating the impact of interventions to control and eliminate malaria. | 2023
  Development and parametrization of mathematical models that incorporate risk heterogeneity in hosts to recapitulate major features of malaria transmission in the study site and estimate the impact of control measures (e.g., insecticide-treated bednet distribution, larviciding or improved antirelapse therapy for vivax malaria).

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo U Ferreira, PhD MD, Study Director — University of Sao Paulo; simone l andrade, Phd MD, Study Chair — Oswaldo Cruz Foundation
Locations (1):
- Marcelo Urbano Ferreira, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johansen IC, Rodrigues PT, Tonini J, Vinetz J, Castro MC, Ferreira MU. Cohort profile: the Mancio Lima cohort study of urban malaria in Amazonian Brazil. BMJ Open. 2021 Nov 17;11(11):e048073. doi: 10.1136/bmjopen-2020-048073. PMID 34789490